CLINICAL TRIAL: NCT02064738
Title: A Pilot Study of the Effectiveness of a High Omega-3/Low Omega-6 Treatment Diet for Treating Aspirin-exacerbated Respiratory Disease
Brief Title: High Omega-3/Low Omega-6 Treatment Diet for Aspirin-exacerbated Respiratory Disease (AERD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Tanya Laidlaw, MD, Assistant Professor of Medicine, Harvard Medical School, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2013-P002683
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: ASA Triad; Asthma, Nasal Polyps, And Aspirin Intolerance
Keywords: Omega-3 fatty acids; Omega-6 fatty acids; aspirin exacerbated respiratory disease; AERD; Samter's Triad; nasal polyp; aspirin; diet; leukotriene
MeSH Terms: conditions — Asthma, Nasal Polyps, And Aspirin Intolerance; Nasal Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal diet (No Intervention): Two weeks of unaltered diet
- Low omega-6/high omega-3 diet (Experimental): Restricting daily intake of omega-6 fatty acids to less than 4 grams and increasing omega-3 fatty acids to 3 grams
  Interventions: Behavioral: Restricting daily intake of omega-6 fatty acids to less than 4 grams and increasing omega-3 fatty acids to 3 grams

INTERVENTIONS:
Behavioral: Restricting daily intake of omega-6 fatty acids to less than 4 grams and increasing omega-3 fatty acids to 3 grams
  Arms: Low omega-6/high omega-3 diet

SUMMARY:
The purpose of this trial is to test the hypothesis that a treatment diet low in omega-6 fatty acids and high in omega-3 fatty acids can cause improvement in asthma symptoms, nasal symptoms, and pulmonary function in patients with aspirin-exacerbated respiratory disease (AERD).

ELIGIBILITY:
Inclusion Criteria:

* History of physician-diagnosed asthma
* History of nasal polyposis
* History of at least two reactions to oral aspirin or other nonselective cyclooxygenase inhibitor with features of lower airway involvement (cough, chest tightness, wheezing, dyspnea), or diagnosis of AERD via a physician-conducted challenge to aspirin
* Age between 18 and 70 years

Exclusion Criteria:

* Current smoking, defined as daily tobacco smoking in the last 6 months and at least one instance of tobacco smoking in the last 3 months.
* Current pregnancy or breastfeeding
* BMI <20
* History of allergy to fish or any unwillingness to eat fish as a regular part of the diet
* Use of Zyflo (zileuton) in the last two weeks
* Presence of an implantable cardioverter-defibrillator
* Use of oral steroids in the last two weeks
* Participation in any other clinical trial in the last month
* Any use of nonsteroidal antiinflammatory drugs (NSAIDs) or any drug that inhibits the cyclooxygenase enzyme during the course of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change in urinary leukotriene E4 levels | 2 weeks and 4 weeks
Change in serum leukotriene B4 levels | 2 weeks and 4 weeks

SECONDARY OUTCOMES:
Change in asthma control questionnaire score | Baseline, 2 weeks, and 4 weeks
Change in Sino-Nasal Outcome Test-22 (SNOT-22) score | Baseline, 2 weeks, and 4 weeks
Change in forced expiratory volume in one second (FEV1), forced vital capacity (FVC), and FEV1/FVC | Baseline, two weeks, and four weeks

OTHER OUTCOMES:
Change in urinary prostaglandin D2 level | 2 weeks and 4 weeks
Change in blood eosinophil count | 2 weeks and 4 weeks
Change in platelet-leukocyte aggregates | 2 weeks and 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tanya M Laidlaw, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: Brigham and Women's Hospital AERD website — http://aerd.partners.org